CLINICAL TRIAL: NCT05739838
Title: Low-Level Laser Effects on Orthodontic Tooth Movement of Periodontally Compromised Patients. Clinical and Biochemical Study
Brief Title: Low-Level Laser Effects on Orthodontic Tooth Movement of Periodontally Compromised Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ORTHO-108-6-J
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Periodontal Diseases; Cancer Metastatic; Orthodontic Tooth Movement
Keywords: Rate of orthodontic tooth movement; Osteiocalsine
MeSH Terms: conditions — Periodontal Diseases; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: ten patients with periodontally affected teeth subjected to low level laser therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontally compromised patients subjected to low level laser therapy (Experimental): periodontally compromised patients with pocket depth of more than 5 mm before receiving nonsurgical periodontal treatment treatment or/and pocket depth of less than 4 mm with periodontal status identified as stable for at least 3 month after nonsurgical periodontal treatment subjected to low-level laser of 940 nm will be applied at day one after start of treatment , weekly during the first month, then monthly.
  Interventions: Device: Biolase ;Low Level Laser
- Periodontally compromised patients (No Intervention): periodontally compromised patients with pocket depth of more than 5 mm before receiving nonsurgical periodontal treatment treatment or/and pocket depth of less than 4 mm with periodontal status identified as stable for at least 3 month after nonsurgical periodontal treatment.

INTERVENTIONS:
Device: Biolase ;Low Level Laser — Low Level laser ,940 nm
  Other Names: Biolase
  Arms: Periodontally compromised patients subjected to low level laser therapy

SUMMARY:
To investigate the effect of Low Level Laser therapy on orthodontic tooth movement of periodontally compromised patients by evaluating the rate of orthodontic tooth movement and the level of Osteocalcin in the gingival crevicular fluid.

DETAILED DESCRIPTION:
Low-Level laser therapy has been reported as an effective adjunct to non surgical periodontal treatment for inflammation control and tissue reparation in patients with periodontitis. Previous studies have shown that application of low-level laser therapy reduced pocket depth and decreased the inflammatory process through regulatory control of inflammatory cytokines level, therefore this study will investigate the effect of low-level laser on the periodontal tissue .Accelerating orthodontic tooth movement is one of the primary demand in orthodontics to prevent side effects as root resorption, caries and decreased patient compliance . Numerous researchers have also studied the use of LLLT in accelerating orthodontic tooth movement and have considered the laser to be effective while others achieved the opposite . Hence, This study is aiming to investigate the effects of LLLT in accelerating tooth movement.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease.
* No history medication (antibiotics and/or anti inflammatory) in the previous 4 months.
* Self motivated patients with acceptable oral hygien.

Exclusion Criteria:

* Previous orthodontic treatment
* Aggressive periodontitis
* Smokers
* pregnant patients

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Rate of orthodontic tooth movement | 6 months
  Rate of mandibular canine retraction

SECONDARY OUTCOMES:
Osteocalcin level in GCF | 6 months
  Gingival Crevicular Fluid samples will be collected from al target teeth in both groups to detect osteocalcin level after start of orthodontic treatment and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Mohsena A Abdelrazek, Lecturer, Study Director — Lecturer of Orthodontic department faculty of Dental medicine for Girls AL-azhar University
Locations (1):
- Faculty of dental medicine for Girls, AL Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Investigate the effect of low level laser on orthodontic tooth movement of periodontally compromised patients, by evaluating the rate of orthodontic tooth movement and the level of osteocalcin in Gingival crevicular fluid

REFERENCES:
- [Background] Ren C, McGrath C, Gu M, Jin L, Zhang C, Sum FHKMH, Wong KWF, Chau ACM, Yang Y. Low-level laser-aided orthodontic treatment of periodontally compromised patients: a randomised controlled trial. Lasers Med Sci. 2020 Apr;35(3):729-739. doi: 10.1007/s10103-019-02923-0. Epub 2019 Dec 12. PMID 31833004